CLINICAL TRIAL: NCT01594242
Title: A Phase 0 Study of Autophagy Induction After Bortezomib For Myeloma
Brief Title: Autophagy Induction After Bortezomib for Myeloma
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 05411
Record Dates: First submitted 2012-04-19; First posted 2012-05-09 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Multiple Myeloma
Keywords: multiple myeloma; bortezomib; proteasome inhibitor
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib

STUDY DESIGN:
Intervention Model Description: Patients who are planned to start a bortezomib-containing regimen (whether for newly diagnosed or relapsed myeloma) will begin with one week off therapy and then one week of single agent bortezomib to allow investigation of its effects on cellular metabolism. Patients may then go on to receive bortezomib in whatever combination is planned by their treating oncologist.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Autophagy Induction After Bortezomib (Experimental): Subjects will undergo a baseline bone marrow aspirate and biopsy (under sedation if preferred by the subject) and have baseline blood samples (and urine samples if clinically indicated for measurement of their myeloma).
  The following week, subjects will undergo a second bone marrow aspirate and biopsy and have additional blood samples taken for research assays prior to starting therapy on treatment day 1 with bortezomib at the standard dose of 1.3 mg/m2. Subjects will receive a second dose of bortezomib on treatment day 4, followed by a third bone marrow aspirate and biopsy on treatment day 4 or 5, along with serial blood samples on treatment days 4 and 5. After completion of the week of study treatment, subjects may continue treatment with the bortezomib-containing regimen planned by their treating oncologist. Active study participation will end after the completion of the week of study treatment.
  Interventions: Drug: Bortezomib

INTERVENTIONS:
Drug: Bortezomib

SUMMARY:
The purpose of this study is to better understand the effects of the chemotherapy medication bortezomib on cancer cells. The investigators are therefore taking blood and bone marrow samples from patients with myeloma who are receiving bortezomib to see if the investigators can detect autophagy in the myeloma cells from the bone marrow and in immune cells in the blood. Subjects are eligible if their doctor is planning to treat them with bortezomib for the first time for their myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

The primary objective of this study is to determine whether administration of bortezomib leads to an increase in cellular autophagy, as determined by electron micrographs of peripheral blood lymphocytes and primary myeloma cells in patients receiving single-agent bortezomib.

SECONDARY OBJECTIVES

1. To determine the optimal timing of autophagy assessments for patients receiving bortezomib.
2. To explore whether high levels of autophagy are associated with resistance to bortezomib therapy.
3. To validate our primary assay by confirming baseline stability of the number of autophagic vesicles per cell
4. To compare results of autophagy measurements in peripheral blood mononuclear cells and bone marrow plasma cells

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed multiple myeloma (both newly diagnosed and relapsed patients are permitted)
* No more than one line of prior therapy containing bortezomib. No prior therapy with any other proteasome inhibitor.
* For subjects who received previous bortezomib, at least a partial response while on the bortezomib-containing therapy, without progression while on bortezomib-containing therapy or within 90 days of stopping bortezomib.
* Planned therapy, as determined by the patient's treating physician, with a bortezomib-containing regimen
* Medically suitable to undergo study procedures, including a one-week washout of prior therapy, one week of observation, and one week of single-agent bortezomib
* Provision of written informed consent

Exclusion Criteria

* Age <18 years (though the demographics of myeloma make it highly unlikely that any children will meet inclusion criteria)
* Treatment with other anti-myeloma agents, including corticosteroids, thalidomide, or lenalidomide, within the 7 days prior to the study baseline bone marrow biopsy.
* Inability to understand the informed consent document or unwillingness to consent.
* Written informed consent must be obtained from all patients before study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2012-07-10 (Actual); Primary Completion 2015-03-02 (Actual); Study Completion 2015-03-02 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Dan Vogl, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States